CLINICAL TRIAL: NCT02328820
Title: DEFINE-FLOW (Distal Evaluation of Functional Performance With Intravascular Sensors to Assess the Narrowing Effect - Combined Pressure and Doppler FLOW Velocity Measurements)
Brief Title: Combined Pressure and Flow Measurements to Guide Treatment of Coronary Stenoses
Acronym: DEFINE-FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Volcano Corporation (Industry)
Responsible Party: Principal Investigator, Nils Johnson, Associate Professor of Medicine, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-14-0442; NL48375.018.14 (Other: Academic Medical Center (AMC), University of Amsterdam)
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve, Myocardial; Coronary Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Other): All lesions undergo simultaneous assessment with a combined pressure and flow sensor
  Interventions: Other: Percutaneous coronary intervention (PCI); Other: Optimal medical therapy (OMT)

INTERVENTIONS:
Other: Percutaneous coronary intervention (PCI) — For lesions with both FFR<=0.8 and CFR<2.0
Other: Optimal medical therapy (OMT) — For lesions with FFR>0.8 or CFR>=2.0 or both

SUMMARY:
This study evaluates the prognostic value and therapeutic potential of combined pressure and flow measurements when evaluating a coronary artery stenosis. Lesions with intact coronary flow reserve (CFR) despite a reduced fractional flow reserve (FFR) will receive optimal medical therapy. Only lesions with a simultaneous reduction in both CFR and FFR will be treated with percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Pressure and flow represent the two physiologic variables that can be measured directly inside a coronary artery. Already pressure measurements have proven their clinical value in the form of fractional flow reserve (FFR). However, myocardial function can remain intact with sufficient flow, even at a low perfusion pressure. Therefore, combined pressure and flow measurements provide a more complete description of physiologic stenosis severity as a guide to medical treatment versus revascularization. Based on existing work relating the most common flow measurement, coronary flow reserve (CFR), to FFR and linking both variables with subsequent prognosis, we hypothesize that lesions with an intact CFR>=2.0 can be reasonably treated with medical therapy despite a reduced FFR<=0.8.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Eligible for PCI based on local practice standards during the current procedure (PCI cannot be staged).
* At least one epicardial stenosis of ≥50% diameter (by visual or quantitative assessment) and meeting the following criteria as determined by the operator based on either a prior or the current diagnostic angiogram:

  * <100% diameter (not a chronic, total occlusion);
  * in a native coronary artery (including side branches but excludes bypass grafts);
  * of ≥2.5mm reference diameter (near the level of the stenosis);
  * and supplies sufficiently viable myocardium (exclude regions of known, prior, transmural myocardial infarction).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Anatomic exclusions:

  * Prior CABG.
  * Preferred treatment strategy for revascularization would be CABG based on local practice standards.
  * Left main coronary artery disease requiring revascularization.
  * Extremely tortuous or calcified coronary arteries precluding intracoronary physiologic measurements. Operators may also exclude subtotal or similar high-grade lesions, which in their judgment may be threatened by ComboWire placement.
  * Known severe LV hypertrophy (septal wall thickness at echocardiography of >13 mm).
* Clinical exclusions:

  * Inability to receive intravenous adenosine (for example, severe reactive airway disease, marked hypotension, or high-grade AV block without pacemaker).
  * Recent (within 3 weeks prior to cardiac catheterization) ST-segment elevation myocardial infarction (STEMI) in any arterial distribution (not specifically target lesion).
  * Culprit lesions (based on clinical judgment of the operator) for either STEMI or non-STEMI cannot be included.
  * Severe cardiomyopathy (LV ejection fraction <30%).
  * Planned need for cardiac surgery (for example, valve surgery, treatment of aortic aneurysm, or septal myomectomy).
* General exclusions:

  * A life expectancy of less than 2 years.
  * Inability to sign an informed consent, due to any mental condition that renders the subject unable to understand the nature, scope, and possible consequences of the trial or due to mental retardation or language barrier.
  * Potential for non-compliance towards the requirements for follow-up visits.
  * Participation or planned participation in another cardiovascular clinical trial before completing the 24 month follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 24 months
  All-cause death, non-fatal myocardial infarction, urgent and elective revascularization

SECONDARY OUTCOMES:
Angina (Canadian Cardiovascular Society (CCS) anginal class (or freedom from angina) | 24 months
  Canadian Cardiovascular Society (CCS) anginal class (or freedom from angina)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Johnson, MD, Principal Investigator — University of Texas Medical School at Houston; Jan J Piek, MD, PhD, Study Director — Academic Medical Center (AMC), Amsterdam
Locations (12):
- Aarhus University Hospital, Aarhus, Denmark
- Catholic University of the Sacred Heart, Rome, Italy
- Japan (4):
  - Gifu Heart Center, Gifu
  - Toda Central General Hospital, Toda
  - Tokyo Medical University, Tokyo
  - Tsuchiura Kyodo, Tsuchiura
- Netherlands (4):
  - Amsterdam UMC - location AMC, Amsterdam
  - Amsterdam UMC - location VUmc, Amsterdam
  - Tergooi Hospital, Blaricum
  - Amphia Hospital, Breda
- Hospital Clinico San Carlos, Madrid, Spain
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Background] Johnson NP, Kirkeeide RL, Gould KL. Is discordance of coronary flow reserve and fractional flow reserve due to methodology or clinically relevant coronary pathophysiology? JACC Cardiovasc Imaging. 2012 Feb;5(2):193-202. doi: 10.1016/j.jcmg.2011.09.020. PMID 22340827
- [Background] van de Hoef TP, van Lavieren MA, Damman P, Delewi R, Piek MA, Chamuleau SA, Voskuil M, Henriques JP, Koch KT, de Winter RJ, Spaan JA, Siebes M, Tijssen JG, Meuwissen M, Piek JJ. Physiological basis and long-term clinical outcome of discordance between fractional flow reserve and coronary flow velocity reserve in coronary stenoses of intermediate severity. Circ Cardiovasc Interv. 2014 Jun;7(3):301-11. doi: 10.1161/CIRCINTERVENTIONS.113.001049. Epub 2014 Apr 29. PMID 24782198
- [Derived] Tas A, Alan Y, Tas IK, Aydin OE, Atay Z, Yilmaz S, Ozcan A, van de Hoef TP, Umman S, Piek Md JJ, Sezer M. Coronary Microvascular Dysfunction Alters the Pulsatile Behavior of the Resting Coronary Blood Flow. Microcirculation. 2025 Aug;32(6):e70021. doi: 10.1111/micc.70021. PMID 40831095
- [Derived] Tas A, Alan Y, Kara Tas I, Umman S, Parker KH, van de Hoef TP, Sezer M, Piek JJ. The impact of high microvascular resistance on coronary wave energetics depends on coronary microvascular functionality. Eur Heart J Open. 2025 May 5;5(3):oeaf050. doi: 10.1093/ehjopen/oeaf050. eCollection 2025 May. PMID 40417173
- [Derived] Tas A, Alan Y, Muftuogullari A, Haj Mohammad AIM, Umman S, Parker KH, Sezer M. Coronary microvascular dysfunction and autoregulatory capacity interfere with resting Dicrotic notch morphology. Microvasc Res. 2025 Jan;157:104750. doi: 10.1016/j.mvr.2024.104750. Epub 2024 Sep 30. PMID 39357645
- [Derived] Achim A, Johnson NP, Liblik K, Burckhardt A, Krivoshei L, Leibundgut G. Coronary steal: how many thieves are out there? Eur Heart J. 2023 Aug 7;44(30):2805-2814. doi: 10.1093/eurheartj/ehad327. PMID 37264699
- [Derived] van de Hoef TP, Stegehuis VE, Madera-Cambero MI, van Royen N, van der Hoeven NW, de Waard GA, Meuwissen M, Christiansen EH, Eftekhari A, Niccoli G, Lockie T, Matsuo H, Nakayama M, Kakuta T, Tanaka N, Casadonte L, Spaan JAE, Siebes M, Tijssen JGP, Escaned J, Piek JJ. Impact of core laboratory assessment on treatment decisions and clinical outcomes using combined fractional flow reserve and coronary flow reserve measurements - DEFINE-FLOW core laboratory sub-study. Int J Cardiol. 2023 Apr 15;377:9-16. doi: 10.1016/j.ijcard.2023.01.009. Epub 2023 Jan 11. PMID 36640965
- [Derived] Eftekhari A, Westra J, Stegehuis V, Holm NR, van de Hoef TP, Kirkeeide RL, Piek JJ, Lance Gould K, Johnson NP, Christiansen EH. Prognostic value of microvascular resistance and its association to fractional flow reserve: a DEFINE-FLOW substudy. Open Heart. 2022 Apr;9(1):e001981. doi: 10.1136/openhrt-2022-001981. PMID 35410913
- [Derived] Johnson NP, Collet C. Can FFR After Stenting Help Reduce Target Vessel Failure? JACC Cardiovasc Interv. 2021 Sep 13;14(17):1901-1903. doi: 10.1016/j.jcin.2021.08.001. No abstract available. PMID 34503740
- [Derived] Murai T, Stegehuis VE, van de Hoef TP, Wijntjens GWM, Hoshino M, Kanaji Y, Sugiyama T, Hamaya R, Nijjer SS, de Waard GA, Echavarria-Pinto M, Knaapen P, Meuwissen M, Davies JE, van Royen N, Escaned J, Siebes M, Kirkeeide RL, Gould KL, Johnson NP, Piek JJ, Kakuta T. Coronary Flow Capacity to Identify Stenosis Associated With Coronary Flow Improvement After Revascularization: A Combined Analysis From DEFINE FLOW and IDEAL. J Am Heart Assoc. 2020 Jul 21;9(14):e016130. doi: 10.1161/JAHA.120.016130. Epub 2020 Jul 14. PMID 32660310
- [Derived] Stegehuis VE, Wijntjens GWM, van de Hoef TP, Casadonte L, Kirkeeide RL, Siebes M, Spaan JAE, Gould KL, Johnson NP, Piek JJ. Distal Evaluation of Functional performance with Intravascular sensors to assess the Narrowing Effect-combined pressure and Doppler FLOW velocity measurements (DEFINE-FLOW) trial: Rationale and trial design. Am Heart J. 2020 Apr;222:139-146. doi: 10.1016/j.ahj.2019.08.018. Epub 2019 Sep 1. PMID 32062172
- [Derived] Gould KL, Johnson NP, Roby AE, Nguyen T, Kirkeeide R, Haynie M, Lai D, Zhu H, Patel MB, Smalling R, Arain S, Balan P, Nguyen T, Estrera A, Sdringola S, Madjid M, Nascimbene A, Loyalka P, Kar B, Gregoric I, Safi H, McPherson D. Regional, Artery-Specific Thresholds of Quantitative Myocardial Perfusion by PET Associated with Reduced Myocardial Infarction and Death After Revascularization in Stable Coronary Artery Disease. J Nucl Med. 2019 Mar;60(3):410-417. doi: 10.2967/jnumed.118.211953. Epub 2018 Aug 16. PMID 30115688
- [Derived] Matsumura M, Johnson NP, Fearon WF, Mintz GS, Stone GW, Oldroyd KG, De Bruyne B, Pijls NHJ, Maehara A, Jeremias A. Accuracy of Fractional Flow Reserve Measurements in Clinical Practice: Observations From a Core Laboratory Analysis. JACC Cardiovasc Interv. 2017 Jul 24;10(14):1392-1401. doi: 10.1016/j.jcin.2017.03.031. PMID 28728652
- [Derived] Johnson NP, Gould KL, Di Carli MF, Taqueti VR. Invasive FFR and Noninvasive CFR in the Evaluation of Ischemia: What Is the Future? J Am Coll Cardiol. 2016 Jun 14;67(23):2772-2788. doi: 10.1016/j.jacc.2016.03.584. PMID 27282899
- [Derived] Gould KL, Johnson NP. Coronary Blood Flow After Acute MI: Alternative Truths. JACC Cardiovasc Interv. 2016 Mar 28;9(6):614-7. doi: 10.1016/j.jcin.2016.02.009. No abstract available. PMID 27013162
- [Derived] Gould KL. Intense Exercise and Native Collateral Function in Stable Moderate Coronary Artery Disease: Incidental, Causal, or Clinically Important? Circulation. 2016 Apr 12;133(15):1431-4. doi: 10.1161/CIRCULATIONAHA.116.022037. Epub 2016 Mar 15. No abstract available. PMID 26979084
- [Derived] Gould KL, Johnson NP. Myocardial Bridges: Lessons in Clinical Coronary Pathophysiology. JACC Cardiovasc Imaging. 2015 Jun;8(6):705-9. doi: 10.1016/j.jcmg.2015.02.013. No abstract available. PMID 26068287
- [Derived] Gould KL, Johnson NP, Kaul S, Kirkeeide RL, Mintz GS, Rentrop KP, Sdringola S, Virmani R, Narula J. Patient selection for elective revascularization to reduce myocardial infarction and mortality: new lessons from randomized trials, coronary physiology, and statistics. Circ Cardiovasc Imaging. 2015 May;8(5):e003099. doi: 10.1161/CIRCIMAGING.114.003099. No abstract available. PMID 25977304